CLINICAL TRIAL: NCT06366685
Title: Development and Initial Application of a Combined Exercise and Psychological Intervention Program for Patients After Esophagectomy
Acronym: Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mengmeng Yuan (Other)
Collaborators: Anhui Medical University (Other)
Responsible Party: Sponsor-Investigator, Mengmeng Yuan, Research Assistant, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: YJS20230170
Record Dates: First submitted 2024-04-06; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Cancer; Exercise Training; Psychotherapy; Rehabilitation
Keywords: Esophageal cancer; Esophagectomy; Rehabilitation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Exercise; Psychosocial Intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise training (Experimental): Implementing only exercise intervention for participants, including aerobic exercise, breathing exercises, resistance exercises, with specific exercise regimes tailored to the participants' physical conditions.
  Interventions: Behavioral: Exercise and Psychological Intervention
- Mindfulness-Based Stress Reduction Therapy (Experimental): Implementing only mindfulness-based stress reduction therapy as the main psychological intervention for participants, and dynamically adjusting based on the participants' psychological states.
  Interventions: Behavioral: Exercise and Psychological Intervention
- Exercise combined with Mindfulness-Based Stress Reduction Therapy (Experimental): Implementing intervention combining exercise with mindfulness-based stress reduction therapy for participants, and dynamically adjusting based on the participants' physical and mental recovery status.
  Interventions: Behavioral: Exercise and Psychological Intervention
- Routine care (No Intervention): Implementing only the department's routine care for esophageal cancer surgical patients.

INTERVENTIONS:
Behavioral: Exercise and Psychological Intervention — To address the symptoms and severity experienced by esophageal cancer patients after surgery, providing them with exercise or psychological interventions to improve their rehabilitation outcomes.
  Arms: Exercise combined with Mindfulness-Based Stress Reduction Therapy; Exercise training; Mindfulness-Based Stress Reduction Therapy

SUMMARY:
Esophageal cancer imposes a significant burden in China, accounting for over 60% of the global disease burden. While surgery remains a common and highly effective treatment for esophageal cancer, patients often experience multiple physical and psychological symptoms postoperatively, severely affecting their recovery outcomes and quality of life. Although existing exercise or psychological intervention programs have shown some effectiveness, issues such as relatively singular intervention content, imprecise intervention timing, and vague intervention details persist.

This project, based on previous research foundations (including the development of symptom measurement tools and the identification of key recovery periods), is guided by symptom management theory and knowledge translation models. Taking a perspective of the synergistic impact of physical and psychological symptoms, the study focuses on patients undergoing esophageal cancer surgery. Initially, evidence-based literature review, focus group interviews, and expert consultations were conducted to develop a combined exercise and psychological intervention program, integrating subjective (CSCA_EC) and objective (6MWT) measurement indicators, named "Recovery For EC." Subsequently, the program was preliminarily applied in clinical settings using a mixed-methods approach, combining quantitative quasi-experimental design (108 cases) and qualitative interviews to assess its acceptability. The final clinical trial version of the Recovery For EC program was developed to provide patients with a tool for self-monitoring recovery outcomes and offer clinical healthcare professionals guidance for implementing precise and personalized rehabilitation management.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of esophageal cancer by pathological biopsy.
2. Undergoing surgical treatment.
3. Age ≥ 18 years old.
4. The patient is able to communicate effectively in language.
5. The patient is fully aware of their condition and willingly participates in the investigation.

Exclusion Criteria:

1. Patients with consciousness disorders.
2. Patients with severe physical illnesses who are unable to cooperate with the investigation.
3. Participation in other studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
the Convalescence Symptom Assessment Scale for EsophageCtomy patients (CSAS_EC) | Preoperative and Postoperative day 7 and through study completion, on average, 40 days post-surgery.
  The Convalescence Symptom Assessment Scale for EsophageCtomy patients (CSAS_EC) is an instrument developed by our research team based on patient self-reported outcomes, designed to assess the symptomatology and functional level during the recovery period of esophagectomy patients. This CSAS_EC has been developed and refined into an 11-point scale with 28 items, encompassing four dimensions (early recovery symptoms, late recovery symptoms, persistent symptoms, and psychosocial symptoms). The CSAS_EC scores range from 0 to 280, with higher scores indicating more severe postoperative symptoms in esophageal cancer patients.

SECONDARY OUTCOMES:
6-Minute Walk Test | Preoperative and Postoperative day 7 and through study completion, on average, 40 days post-surgery.
  Participants are instructed to walk as fast as possible in a sparsely crowded, straight corridor to determine their six-minute walking distance. The cardiorespiratory functional assessment criteria are as follows: walking distance <150 meters is considered severely abnormal, 150-300 meters is moderately abnormal, 301-450 meters is mildly abnormal, and >450 meters is considered normal.
Hospital Anxiety and Depression Scale (HADS) | Preoperative and Postoperative day 7 and through study completion, on average, 40 days post-surgery.
  The Hospital Anxiety and Depression Scale (HADS) is a widely used self-assessment questionnaire for evaluating anxiety and depression symptoms in hospital patients. HADS consists of 14 items, divided into two dimensions: Anxiety and Depression. It uses a Likert 4-point scale, with scores ranging from 0 to 21. Higher scores indicate more severe anxiety and depression symptoms.
Postoperative Complications | Postoperative day 7
  According to the Clavien-Dindo classification system, Grade I refers to complications that do not require any treatment such as medication or surgery, Grade II involves the need for medication, blood transfusion, or nutritional support, Grade III necessitates surgical or interventional treatment, Grade IV poses a potential threat to the patient's life requiring intensive care, and Grade V results in patient death. The number and severity of postoperative complications are assessed and documented accordingly. Data on complications can be obtained from participants' electronic medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes
The plan includes sharing raw data, which requires approval from the corresponding author of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Access to the relevant data at the conclusion of this study is permitted, and its usage may be determined based on the needs of the user, subject to approval from the corresponding author of the study.
Access Criteria: Approval from the corresponding author of the study is required.

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Liu CQ, Ma YL, Qin Q, Wang PH, Luo Y, Xu PF, Cui Y. Epidemiology of esophageal cancer in 2020 and projections to 2030 and 2040. Thorac Cancer. 2023 Jan;14(1):3-11. doi: 10.1111/1759-7714.14745. Epub 2022 Dec 8. PMID 36482832
- [Result] Ma X, Ge H, Zhang X, Li S. Survival experience of patients undergoing oesophagectomy during the recovery period: A meta-synthesis of qualitative studies. J Clin Nurs. 2023 Sep;32(17-18):5579-5595. doi: 10.1111/jocn.16648. Epub 2023 Feb 17. PMID 36802111
- [Result] Liu L, Liu QW, Wu XD, Liu SY, Cao HJ, Hong YT, Qin HY. Follow-up study on symptom distress in esophageal cancer patients undergoing repeated dilation. World J Clin Cases. 2020 Aug 26;8(16):3503-3514. doi: 10.12998/wjcc.v8.i16.3503. PMID 32913857
- [Result] Gupta V, Allen-Ayodabo C, Davis L, Zhao H, Hallet J, Mahar AL, Ringash J, Kidane B, Darling G, Coburn NG. Patient-Reported Symptoms for Esophageal Cancer Patients Undergoing Curative Intent Treatment. Ann Thorac Surg. 2020 Feb;109(2):367-374. doi: 10.1016/j.athoracsur.2019.08.030. Epub 2019 Sep 21. PMID 31550465
- [Result] Hellstadius Y, Lagergren P, Lagergren J, Johar A, Hultman CM, Wikman A. Aspects of emotional functioning following oesophageal cancer surgery in a population-based cohort study. Psychooncology. 2015 Jan;24(1):47-53. doi: 10.1002/pon.3583. Epub 2014 Jun 3. PMID 24895142
- [Result] Ohkura Y, Ichikura K, Shindoh J, Ueno M, Udagawa H, Matsushima E. Association between psychological distress of each points of the treatment of esophageal cancer and stress coping strategy. BMC Psychol. 2022 Sep 6;10(1):214. doi: 10.1186/s40359-022-00914-5. PMID 36068609
- [Result] Liu Y, Pettersson E, Schandl A, Markar S, Johar A, Lagergren P. Psychological distress after esophageal cancer surgery and the predictive effect of dispositional optimism: a nationwide population-based longitudinal study. Support Care Cancer. 2022 Feb;30(2):1315-1322. doi: 10.1007/s00520-021-06517-x. Epub 2021 Sep 4. PMID 34480622
- [Result] Johns SA, Von Ah D, Brown LF, Beck-Coon K, Talib TL, Alyea JM, Monahan PO, Tong Y, Wilhelm L, Giesler RB. Randomized controlled pilot trial of mindfulness-based stress reduction for breast and colorectal cancer survivors: effects on cancer-related cognitive impairment. J Cancer Surviv. 2016 Jun;10(3):437-48. doi: 10.1007/s11764-015-0494-3. Epub 2015 Nov 19. PMID 26586494
- [Result] Lee JY, Park HY, Jung D, Moon M, Keam B, Hahm BJ. Effect of brief psychoeducation using a tablet PC on distress and quality of life in cancer patients undergoing chemotherapy: a pilot study. Psychooncology. 2014 Aug;23(8):928-35. doi: 10.1002/pon.3503. Epub 2014 Feb 18. PMID 24535848
- [Result] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Result] Anandavadivelan P, Malberg K, Vikstrom K, Nielsen S, Holdar U, Johar A, Lagergren P. Home-based physical activity after treatment for esophageal cancer-A randomized controlled trial. Cancer Med. 2023 Feb;12(3):3477-3487. doi: 10.1002/cam4.5131. Epub 2022 Aug 18. PMID 36812121
- [Result] van Vulpen JK, Hiensch AE, van Hillegersberg R, Ruurda JP, Backx FJG, Nieuwenhuijzen GAP, Kouwenhoven EA, Groenendijk RPR, van der Peet DL, Hazebroek EJ, Rosman C, Wijnhoven BPL, van Berge Henegouwen MI, van Laarhoven HWM, Siersema PD, May AM. Supervised exercise after oesophageal cancer surgery: the PERFECT multicentre randomized clinical trial. Br J Surg. 2021 Jul 23;108(7):786-796. doi: 10.1093/bjs/znab078. PMID 33837380
- [Result] Hofmann SG, Gomez AF. Mindfulness-Based Interventions for Anxiety and Depression. Psychiatr Clin North Am. 2017 Dec;40(4):739-749. doi: 10.1016/j.psc.2017.08.008. Epub 2017 Sep 18. PMID 29080597
- [Result] Chinh K, Mosher CE, Brown LF, Beck-Coon KA, Kroenke K, Johns SA. Psychological Processes and Symptom Outcomes in Mindfulness-Based Stress Reduction for Cancer Survivors: A Pilot Study. Mindfulness (N Y). 2020 Apr;11(4):905-916. doi: 10.1007/s12671-019-01299-0. Epub 2020 Jan 14. PMID 33456623
- [Result] Victorson D, Murphy K, Benedict C, Horowitz B, Maletich C, Cordero E, Salsman JM, Smith K, Sanford S. A randomized pilot study of mindfulness-based stress reduction in a young adult cancer sample: Feasibility, acceptability, and changes in patient reported outcomes. Psychooncology. 2020 May;29(5):841-850. doi: 10.1002/pon.5355. Epub 2020 Feb 25. PMID 32040222